CLINICAL TRIAL: NCT02391298
Title: An Examination of Potential Neurochemical and Cognitive Mediators of the Relationship Between Mindfulness and Emotion Regulation in Individuals With Multiple Sclerosis: An Internet Based Self-Guided Pilot Study.
Brief Title: An Online Self-Guided Meditation Course for Individuals With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haley Duncanson (Other)
Collaborators: Suffolk University (Other)
Responsible Party: Sponsor-Investigator, Haley Duncanson, Co-Investigator, Suffolk University
Organization: Suffolk University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SuffolkU
Record Dates: First submitted 2015-03-08; First posted 2015-03-18 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; stress; meditation; attention
MeSH Terms: conditions — Multiple Sclerosis | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mindfulness Meditation (Experimental): All participants will complete baseline assessments of variables of interest (i.e., levels of mindfulness, contrast sensitivity, cognitive inhibition, and emotional regulation skills). Participants will then undergo 8 weeks of self-directed mindfulness training with re-assessments of variables of interest completed at week 4 and week 8. All participants will be given access to meditation recordings and asked to practice the exercises in a progressive manner from mindfulness of breath to a loving/kindness meditation (each exercise twice per week). Participants will be asked at the end of study for feedback on the acceptability of the program.
  Interventions: Behavioral: Mindfulness Meditation

INTERVENTIONS:
Behavioral: Mindfulness Meditation

SUMMARY:
The aim of this study is to examine whether meditation delivered by the internet improves mood and attention as well as increases levels of dopamine in individuals who have been diagnosed with Multiple Sclerosis.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is thought to involve a chronic, autoimmune inflammatory process in which one's own immune system attacks the myelin sheath surrounding axons in the central nervous system. MS is associated with many symptoms that decrease one's quality of life including pain, spasticity, fatigue, bowel and bladder problems, dizziness, cognitive difficulties, and depression. There is currently no cure for MS.

Decreased levels of dopamine (DA) have been measured in the cerebrospinal fluid of those with the primary progressive type of MS. In individuals with the relapsing- remitting type of MS, dopamine levels showed a negative correlation to disease severity such that as dopamine levels decreased, disease severity increased. Additionally, many symptoms of MS are related to dopaminergic dysfunction and/or abnormalities in dopamine rich brain areas. Dopamine levels have been shown to increase via active meditation during PET imaging in long term meditators. Other studies have also linked dopamine release to meditation in the peripheral nervous system (via measures of a DA metabolite in blood plasma levels). It is not clear whether brief meditation training in naive participants may have similar effects. Whether meditation could enhance dopamine levels in patients with MS or meditation naïve individuals has not been studied. Both dopamine and mindfulness training have been linked to improved attention and emotion regulation. Research has also indicated that attentional failures and infrequent use of emotion regulation strategies predicted poorer quality of life in patients with MS. Thus, there is sufficient evidence to suggest that meditation can enhance attention, emotion regulation, and quality of life in individuals with MS and that dopamine may be a neurochemical mechanism for this change.

This study is an open trial pilot design with multiple assessments on measures of mindfulness, dopamine, inhibition, and emotion regulation. The primary goal of the current study is evaluate the efficacy of an internet based mindfulness program for individuals with MS. The investigators hypothesize that individuals with MS will show increased levels of mindfulness and improved emotion regulation and cognitive inhibition skills after the course. In addition, The investigators hypothesize that contrast sensitivity (a proxy measure of retinal dopamine levels) will increase after the course. A secondary goal of this study is to examine potential cognitive and neurochemical mechanisms of mindfulness in relation to emotion regulation. Specifically, the investigators propose to examine whether dopamine and cognitive inhibition mediate the relationship between mindfulness and improved emotion regulation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis
* Must be available for 2 in person visits in Massachusetts

Exclusion Criteria:

* Patients with psychosis.
* Self-reported disorders of the central nervous system other than MS.
* Participants currently engaged in weekly psychotherapy who are unable to reduce session to once per month for the duration of the study.
* Sensorimotor limitations that would confound test results.
* Daily meditation practice (current or during the last 3 months).
* Medication changes in the past 3 months.
* Participants who, due to their MS are medically unstable. This will be defined as anyone who is actively relapsing at the time of recruitment (or within the last two weeks), or who becomes symptomatic during training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The Stop Signal Test (SST) | Change from baseline of total correct responses on SST at 8 weeks
  Measure of Cognitive Inhibition
The Freiburg Visual Acuity Test (FrACT) | Change from baseline of contrast sensitivity at 8 weeks
  Measure of Contrast Sensitivity

SECONDARY OUTCOMES:
The Functional Assessment of Multiple Sclerosis (FAMS) Quality of Life Instrument | Baseline and 8 weeks
  self-report scale that assesses a range aspects of quality of life reported to be important by individuals with MS.
Feedback Questionnaire | 8 weeks
  This self-report questionnaire was created in order to gather information regarding feasibility, acceptability, and general impressions of the program from participants.
Mindful Attention Awareness Scale | Change from baseline in mindfulness skills at 8 weeks
  Self-report measure of levels of mindfulness
Difficulties in Emotion Regulation Scale | Change from baseline in emotion regulation skills at 8 weeks
  self-report measure of emotional regulation skills

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Moes, PhD, Principal Investigator — Suffolk University
Locations (1):
- Suffolk University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Logan GD, Cowan WB, Davis KA. On the ability to inhibit simple and choice reaction time responses: a model and a method. J Exp Psychol Hum Percept Perform. 1984 Apr;10(2):276-91. doi: 10.1037//0096-1523.10.2.276. PMID 6232345
- [Background] Verbruggen F, Logan GD, Stevens MA. STOP-IT: Windows executable software for the stop-signal paradigm. Behav Res Methods. 2008 May;40(2):479-83. doi: 10.3758/brm.40.2.479. PMID 18522058
- [Background] Bach M. The Freiburg Visual Acuity test--automatic measurement of visual acuity. Optom Vis Sci. 1996 Jan;73(1):49-53. doi: 10.1097/00006324-199601000-00008. PMID 8867682
- [Background] Cella DF, Dineen K, Arnason B, Reder A, Webster KA, karabatsos G, Chang C, Lloyd S, Steward J, Stefoski D. Validation of the functional assessment of multiple sclerosis quality of life instrument. Neurology. 1996 Jul;47(1):129-39. doi: 10.1212/wnl.47.1.129. PMID 8710066
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Gratz, K. L., & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of Psychopathology and Behavioral Assessment, 26(1), 41-54.
- [Background] Markianos M, Koutsis G, Evangelopoulos ME, Mandellos D, Karahalios G, Sfagos C. Relationship of CSF neurotransmitter metabolite levels to disease severity and disability in multiple sclerosis. J Neurochem. 2009 Jan;108(1):158-64. doi: 10.1111/j.1471-4159.2008.05750.x. Epub 2008 Nov 12. PMID 19014375
- [Background] Kjaer TW, Bertelsen C, Piccini P, Brooks D, Alving J, Lou HC. Increased dopamine tone during meditation-induced change of consciousness. Brain Res Cogn Brain Res. 2002 Apr;13(2):255-9. doi: 10.1016/s0926-6410(01)00106-9. PMID 11958969
- [Background] Jung YH, Kang DH, Byun MS, Shim G, Kwon SJ, Jang GE, Lee US, An SC, Jang JH, Kwon JS. Influence of brain-derived neurotrophic factor and catechol O-methyl transferase polymorphisms on effects of meditation on plasma catecholamines and stress. Stress. 2012 Jan;15(1):97-104. doi: 10.3109/10253890.2011.592880. Epub 2011 Jul 26. PMID 21790467
- [Background] Jung YH, Kang DH, Jang JH, Park HY, Byun MS, Kwon SJ, Jang GE, Lee US, An SC, Kwon JS. The effects of mind-body training on stress reduction, positive affect, and plasma catecholamines. Neurosci Lett. 2010 Jul 26;479(2):138-42. doi: 10.1016/j.neulet.2010.05.048. Epub 2010 May 28. PMID 20546836
- [Background] Phillips LH, Saldias A, McCarrey A, Henry JD, Scott C, Summers F, Whyte M. Attentional lapses, emotional regulation and quality of life in multiple sclerosis. Br J Clin Psychol. 2009 Mar;48(Pt 1):101-6. doi: 10.1348/014466508X379566. Epub 2008 Nov 26. PMID 19040791